CLINICAL TRIAL: NCT00134225
Title: Multi-Center, Multi-National Study to Demonstrate That Muscle Pattern Recognition is a Reliable and Valid Evaluation Tool for Patients Who Present With Acute, Sub-Acute, or Chronic Symptoms of Neck or Back Pain of a Musculoskeletal Origin
Brief Title: Study to Demonstrate That Muscle Pattern Recognition (MPR) is an Effective Evaluation Tool for Musculoskeletal Neck or Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: iTech Medical, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IMS MPR 480
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2005-10-26 (Estimated); Status verified 2005-08

CONDITIONS: Neck Pain; Low Back Pain
Keywords: Musculoskeletal abnormality; Musculoskeletal physiology; Musculoskeletal disease; Musculoskeletal dysfunction
MeSH Terms: conditions — Neck Pain; Low Back Pain; Musculoskeletal Abnormalities; Musculoskeletal Diseases

INTERVENTIONS:
Device: Muscle Pattern Recognition (MPR)

SUMMARY:
The investigators hypothesize that non able-bodied participants with reported acute, sub-acute, or chronic symptoms of neck or back pain of a musculoskeletal origin will have magnetic resonance imaging (MRI), X-ray and blood parameters that do not demonstrate a statistical difference between "normal" (able-bodied) volunteers.

Muscle pattern recognition (MPR) testing will show statistically different results between these groups. This statistically significant finding in MPR results will enhance a clinician's determination of clinical normality or abnormality.

If this hypothesis is demonstrated, the MPR modality will be the first quantitative tool developed for assisting in the diagnosis of the presence or absence of a musculoskeletal dysfunction in a patient population. The availability of such an evaluation tool to a healthcare provider for patients with soft tissue, non-surgical neck or back complaints will substantially improve the accuracy of diagnosis and case management decisions.

DETAILED DESCRIPTION:
Investigators aim to use data from both the able-bodied and non able-bodied samples to create a normative database for this technology. The primary objective of populating a normative database will be to construct a reliable and valid normative database representative of the North American population for use with a discriminative analysis tool which will differentiate abnormal musculoskeletal function from normal musculoskeletal function.

Study Population: The study population will be composed of 480 asymptomatic participants (able-bodied individuals) and symptomatic (non able-bodied individuals: individuals with musculoskeletal, non-surgical injuries of the neck and back) selected first on the basis of a screening questionnaire.

Upon signing an informed consent to participate in the study, participants will complete screening questionnaires. They will be independently evaluated by two clinicians, well experienced in the field of musculoskeletal medicine, who obtain a detailed medical history with particular attention to the strict inclusion/exclusion criteria and perform a standardized physical examination. This standardized clinical examination consists of the most current "Gold Standard".

Most patients presenting with musculoskeletal complaints of the back or neck and are frequently given this diagnosis solely on the basis of the "first line" healthcare providers' history and physical examinations.

To ensure the statistical strength of the history and physical selection process for further inclusion into the study, participants will undergo two separate clinical examinations. Each will be performed independently by physicians who are specialists in two different fields of practice that commonly see neck and back pain patients and who must agree if a subject is clinically normal or not.

If selected for continued participation, each participant will undergo Magnetic Resonance Imaging (MRI) of the spine (sagittal views of the entire spine), plain X-rays of the entire spine (A/P and Lateral views), blood studies (CBC, Sedimentation Rate, CPK, Calcium, Phosphorous, Pregnancy test, drug screen) and MPR testing.

A total of 480 clinically and lab normal able-bodied/not-able bodied individuals will be selected and examined over a period of twelve months at 4 different centers.

Able-Bodied Participants:

A total of approximately 240 able-bodied participants will be divided by gender (male, female) and by age classes: specifically [18-30 years], [31-45 years], and [46-62 years]. This sample size was selected, in part, because Edgerton et al. reported that recruitment patterns of the neck or back differ dependent upon gender and our goal is to have a population of approximately 120 males and 120 females.

At the close of the study, investigators will segment the population into the three age groups mentioned, the proposed sample sizes are thought to be appropriate for statistical analysis while still capturing a variety of subject types. The overall age range was chosen to represent the main working population in North America, but to not exceed an upper age range where muscle recruitment patterns may vary on a natural evolutionary basis.

The total number of normal/able-bodied participants will be collected from 4 independent research centers in the U.S. and Canada with an expected maximum of approximately 60 individuals per center. A sub-group of 32 randomly assigned able-bodied volunteers will be scheduled for a second MPR test approximately 7 days after their initial testing to examine the reliability of the MPR evaluation tool. In the selection process, every effort will be made to avoid bias toward a non-working population (i.e. testing only in the morning or afternoon) and to obtain representative proportions of the age and race classes existing in North America.

Not Able-Bodied Participants:

Investigators aim to construct a valid and reliable profile of clinically not normal individuals diagnosed as suffering from musculoskeletal neck or back pain that will be used to confirm our hypothesis and the ability of the MPR evaluation to provide valid, reliable, and objective information for the clinician.

These 240 not able-bodied volunteers will be selected using the same inclusion/exclusion criteria and standardized medical histories and physical examinations as above. One exception to the exclusion criteria is that if a not-normal participant uses ongoing medications for control of discomfort, it will be left to the discretion of each investigator as to how that individual's medication profile may affect their pain reporting, physical performance, or compliance with the protocol steps. A 3-day medication "wash-out" will be allowed (and encouraged) if there is any concern about a participant's performance.

In order to conduct an appropriate discriminate analysis, half of the recruited participants will be an able-bodied sample of participants. Half of the participants will fall into the not able-bodied participant sample. Every effort will be made in the selection process to avoid bias toward a non-working population (i.e. testing only in the morning or afternoon) and obtain representative proportions of the age and race classes existing in North America.

During the data collection process, other clinical categories could be defined for additional statistical analysis such as the loci of symptoms (i.e. lumbar, thoracic, cervical), the level of symptoms (lower, mid, or upper back) and the laterality of symptoms (left or right). Upon analysis of the laboratory and image findings (MRI, X-ray, blood tests) other anatomic findings or variations such as degenerative disc disease, size of possible disc protrusions, Sedimentation Rate or CPK values, Schmorld's nodes, etc. may also be discussed.

Not able-bodied volunteers may have long standing back or neck pain or pain symptoms as recently as several days after a date of injury. This more immediate window of pain will be allowed to include acute events but not until or unless the individual is able to perform the nine movements necessary for the MPR testing procedure. The outer time duration of pain was chosen to include individuals with more chronic complaints, but not if other compensatory or secondary gain issues appear present such as may occur with Worker's Compensation claims, disability claims, or litigation. It is the desire of investigators to include appropriate acute, sub-acute, and chronic neck or back pain sufferers.

We believe that the design of this study will prove that the evaluation provided by the MPR testing modality should be the tool of choice for the objective evaluation and case management of patients presenting with musculoskeletal, non-surgical neck and back pain as it will differentiate "normal" (asymptomatic, able-bodied) individuals from those individuals ("not normal") with underlying biomechanical dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

Individuals may participate in this study if they meet the following criteria:

* 18-62 years of age; male or female.
* 4 foot 10 inches to 6 foot 5 inches in height
* No prior back or neck surgery, or structural deformity of the spine
* No orthopedic injury/illness/surgery limiting range of motion of the shoulders
* No ongoing treatments for back or neck pain/injury from a health professional in the last two years.
* No prior loss of work time due to a neck or back injury/illness
* Laboratory studies: complete blood count (CBC); sedimentation rate; creatinine phosphokinase (CPK); calcium; phosphorus; pregnancy test if female; and drug screen. Laboratory studies will be examined by a physician investigator to determine if the findings will exclude the participant from participating successfully in study activities. A positive pregnancy test or drug screen will automatically exclude the participant from the study.
* Clinical examination of the neck and back by two physicians in agreement that the participant may participate in the study.
* Absence of congenital or acquired neuromuscular disease or dysfunction

Exclusion Criteria:

Individuals may not participate in this study if they meet the following criteria:

* Claustrophobia or anxiety associated with being enclosed in narrow spaces
* Muscle weakness or sensory feedback abnormalities that affect(s) gait
* Pregnancy
* Concurrent serious medical illness such as cancer; recent heart attack or stroke; heart rhythm disturbance requiring a pacemaker; diabetes that causes pain; numbness; or decreased circulation in the legs.
* Alcohol or illicit drug abuse.
* History of (or concurrent) psychiatric illness necessitating ongoing "talk" therapy and/or psychotropic medications
* History of back or neck pain lasting more than 3 days or requiring time off of work AND healthcare provider treatments within the last 2 years
* Involved in a lawsuit or receiving worker's compensation or disability payments
* Individuals with pacemakers or pacemaker wires; aneurysm clips; or metallic foreign bodies or metal shavings in the body.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480
Dates: Start 2005-04; Study Completion 2006-12

PRIMARY OUTCOMES:
This study will demonstrate differences in muscle recruitment patterns between individuals who are "normal" (asymptomatic, able-bodied) from those individuals ("not normal") with underlying biomechanical dysfunction of the neck and back

CONTACTS AND LOCATIONS:
Overall Officials: Alan Goldman, MD, Study Director — Impact Medical Solutions, Inc.
Locations (4):
- United States (3):
  - Department of Neurology - UC Irvine, Irvine, California
  - Midwest Consultants for Clinical Trials LLC, Portage, Michigan
  - Advance Clinical Research, Salt Lake City, Utah
- Institute de Rescherche in Physiatrie du Quebec, Montreal, Quebec, Canada

REFERENCES:
- [Background] VR Edgerton, SL Wolf, DJ Levendowski, RI Jenrich, RR Roy (1997). EMG activity in neck and back muscles during selected static postures in adult males and females. Physiology theory and practice. 13:179-195.
- [Background] VR Edgerton, SL Wolf, DJ Levendowski, RL Roy (1996). Evaluating Patterns of EMG Amplitudes for Trunk and Neck Muscles of Patients and Controls. International Journal of Rehabilitation and Health, 2(1).
- [Result] V.R. Edgerton, S.T. Wolf, D.J. Levendowski, and R.R. Roy (1996). Evaluating Patterns of EMG Amplitudes for Back and Trunk Muscles of Patients and Controls. International Journal of Rehabilitation and Health, 2(1).
- [Result] Edgerton VR, Wolf SL, Levendowski DJ, Roy RR. Theoretical basis for patterning EMG amplitudes to assess muscle dysfunction. Med Sci Sports Exerc. 1996 Jun;28(6):744-51. doi: 10.1097/00005768-199606000-00013. PMID 8784762